CLINICAL TRIAL: NCT00028860
Title: A Phase II Trial Of Adjuvant Chemotherapy For High Risk Transitional Cell Carcinoma Of The Urothelium
Brief Title: Combination Chemotherapy Following Surgery in Treating Patients With Urinary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TULCC-RM-002; CDR0000069142 (Registry Identifier: PDQ (Physician Data Query)); AMGEN-TULCC-RM-002; BMS-TULCC-RM-002
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2004-08

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; localized transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Carboplatin; Gemcitabine; Ifosfamide; Paclitaxel; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: ifosfamide
Drug: paclitaxel
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy following surgery in treating patients who have urinary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to treatment failure and disease-free survival in patients with high-risk transitional cell carcinoma of the urothelium treated with adjuvant paclitaxel, ifosfamide, carboplatin, and gemcitabine.
* Determine the tolerability and feasibility of this regimen in these patients.

OUTLINE: Patients are stratified according to disease stage.

Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 1 hour on day 1, ifosfamide IV over 1 hour on days 1-3, and filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 4 and continuing until blood counts recover. Treatment repeats every 21 days for a total of 2 courses.

Beginning 3 weeks after the completion of the second course of chemotherapy, patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 1 hour on day 1. Patients also receive G-CSF SC once daily on days 2-6 and again beginning on day 9 and continuing until blood counts recover. Treatment repeats every 21 days for a total of 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 months, every 6 months for 2 years, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 10-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of transitional cell carcinoma of the urothelium including bladder, ureter, and renal pelvis

  * T3b-4, N0, M0 OR
  * Any T, N1-3, M0
* Cystectomy within the past 8 weeks

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 months

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than ULN
* Albumin no greater than ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy except curatively treated carcinoma in situ of the cervix or non-melanoma skin cancer
* No active serious infection, other serious underlying medical condition, dementia, or significantly altered mental status that would preclude study participation
* No known hypersensitivity to Cremophor EL
* No pre-existing clinically significant grade 2 or greater neuropathy
* No AIDS (HIV positivity alone allowed)
* No known hypersensitivity to E. coli-derived products

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for malignancy
* No neoadjuvant chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for malignancy

Surgery:

* See Disease Characteristics

Other:

* No other concurrent investigational therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-10; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja Mudad, MD, FACP, Study Chair — Tulane University Health Sciences Center
Locations (1):
- Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana, United States